CLINICAL TRIAL: NCT06551610
Title: A Step-Wedged Cluster Randomized Registry-Based Multi-Centre Trial to Compare the Efficacy Between the Canadian TAVI Triage Tool and Standard of Care in TAVI Patients in Ontario, Canada
Brief Title: CAN3T - Canadian TAVI Triage Tool
Acronym: CAN3T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CTO-4926
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; TAVI; Trans-catheter Aortic Valve Implantation; cardiovascular disease; Surgical Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Step-Wedged Cluster Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Triage tool (Active Comparator)
  Interventions: Other: Triage Tool

INTERVENTIONS:
Other: Triage Tool — Tool that uses patient characteristics to triage patients for an earlier procedure date vs the standard of care 12 week wait for procedure.
  Arms: Triage tool

SUMMARY:
The goal of this trial is to see if a tool that may reduce wait times will reduce bad outcomes in participants on the TAVI waitlist. The main questions it aims to answer are:

* How many deaths, hospitalizations, or urgent TAVI procedures take place while participants wait
* Days alive and out of hospital at 30 days and 12 weeks, total health care costs, and wait times

Researchers will compare usual wait times to see if the tool reduces death, hospitalizations, and urgent procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for TAVI who are 18 years or older at one of 11 TAVI hospitals

Exclusion Criteria:

* Any inpatient referrals who have an urgent inpatient TAVI on the same admission
* Any referral during the 1-month transition period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5060 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of using the CAN3T tool in triage compared to standard care, in TAVI patients, including: reduce wait-time adverse events, improve patient-centred outcomes, and reduce wait-time health care utilization. | From the beginning of enrollment and continuing for 32 months.
  Composite of death, all-cause hospitalization or urgent TAVI (in-hospital and unplanned TAVI) on the TAVI waitlist. The waitlist period is defined as period between TAVI referral and first of either death, TAVI procedure or off list.

IPD SHARING:
Plan to Share IPD: No
No personal information or personal health information is being collected from participants.